CLINICAL TRIAL: NCT02541786
Title: Comparison of Dexlansoprazole-based Triple and Rabeprazole-based Triple Therapies for Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, DENG-CHYANG WU, Clinical Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaohsiungMUH
Record Dates: First submitted 2015-08-27; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: dexlansoprazole MR; rabeprazole; Helicobacter pylori; triple therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexlansoprazole based triple therapy (Active Comparator): dexlansoprazole MR 60 mg once daily, clarithromycin 500 mg twice daily, and amoxicillin 1 g twice daily for 7 days
  Interventions: Drug: dexlansoprazole based triple therapy
- rabeprazole-based triple therapy (Experimental): rabeprazole 20 mg twice daily, clarithromycin 500 mg twice daily, and amoxicillin 1 g twice daily for 7 days
  Interventions: Drug: rabeprazole-based triple therapy

INTERVENTIONS:
Drug: dexlansoprazole based triple therapy — dexlansoprazole MR 60 mg once daily+clarithromycin 500 mg twice daily+ amoxicillin 1 g twice daily for 7 days
  Other Names: Dexilant-based triple therapy
  Arms: dexlansoprazole based triple therapy
Drug: rabeprazole-based triple therapy — rabeprazole 20 mg twice daily + clarithromycin 500 mg twice daily + amoxicillin 1 g twice daily for 7 days
  Other Names: Pariet-based triple therapy
  Arms: rabeprazole-based triple therapy

SUMMARY:
Dexlansoprazole MR is the R-enantiomer of lansoprazole that is delivered by a dual delayed release formulation. It is effective for symptom control of patients with gastroesophageal reflux disease. However, its efficacy in the treatment of H.pylori infection remains unclear. This study was conducted to investigate whether the efficacy of single-dose dexlansoprazole MR-based triple therapy was non-inferior to double-dose rabeprazole-based triple therapy in the treatment of H.pylori infection.

DETAILED DESCRIPTION:
Helicobacter pylori (H.pylori) infect more than 50% of humans globally. It is the major cause of chronic gastritis, gastric ulcer, duodenal ulcer, gastric adenocarcinoma and gastric mucosa-associated lymphoid tissue lymphoma (MALToma). H.pylori eradication has become the standard and most widely adopted therapy to cure peptic ulcer disease. This therapy is also strongly recommended in the treatment of H pylori-related MALToma. In regions with high incidence of gastric adenocarcinoma, eradication of H pylori is advocated as a preventative measure. Proton pump inhibitor (PPI) is one of the key medicines in anti-H pylori regimens. It possesses anti-H pylori activity, and, by reducing gastric acid secretion, it also increases bioavailability and activity of some antibiotics. This study was conducted to investigate whether the efficacy of single-dose dexlansoprazole MR-based triple therapy was non-inferior to double-dose rabeprazole-based triple therapy in the treatment of H pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged more than 20 years.
2. H. pylori-infected outpatients
3. Mental and legal ability to give a written informed consent.

Exclusion Criteria:

1. previous H pylori-eradication therapy,
2. ingestion of antibiotics or bismuth within the prior 4 weeks,
3. patients with allergic history to the medications used,
4. patients with previous gastric surgery,
5. the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia),
6. pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The rate of H.pylori eradication | 6 weeks after finishing study drugs
  Evaluate eradication outcome by 13C urea breath test

SECONDARY OUTCOMES:
Drug Compliance | 6 weeks after finishing study drugs
  Good drug compliance measured by number of subjects taking >= 80% eradication medicines

CONTACTS AND LOCATIONS:
Overall Officials: DENG-CHYANG WU, MD, PHD, Study Chair — Kaohsiung Medical University
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City